CLINICAL TRIAL: NCT00005721
Title: Retaining Donors and Increasing Donation Frequency
Status: Completed | Type: Observational
Sponsor: Bloodworks (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4930; R18HL045265 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Blood Donors

SUMMARY:
To retain individuals as blood donors once they have entered the voluntary blood donation system and to increase the frequency of their donations.

DETAILED DESCRIPTION:
BACKGROUND:

The study continued research previously funded as part of a National Research and Demonstration Center (NRDC) in Transfusion Medicine.

DESIGN NARRATIVE:

There were six components to the study. The first identified significant factors influencing regular blood donations by individuals with different donation histories - first-time, second-time, committed (frequent), and lapsed donors. The second component developed and assessed the validity of behavioral models to increase donor retention and to predict whether first and second time donors would contribute again. The third developed donor-retention interventions, especially for the first and second time donors. The fourth component identified homogeneous subgroups among first, second and committed donors who might be receptive to different types of intervention strategies to increase the frequency of their donations. The fifth component evaluated the success of cost-effectiveness of the new interventions compared to existing blood center maintenance strategies. The sixth identified whether or not donors had a limit or ceiling on how often they donated per year.

The investigators drew on two related social psychological theories to combine cognitive and behavioral approaches to blood donor retention and to use the findings to construct a multiattribute model of donor decision-making. A behavioral decision model was used to predict donor behavior prospectively and to target and direct the design of interventions to increase donor retention and the frequency of donations.

Approximately 33 percent of the total project supported the subproject on retaining donors.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Primary Completion 1993-12 (Actual); Study Completion 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Bier — Bloodworks

REFERENCES:
- [Background] Meyer D, Bolgiano DC, Sayers M, Price T, Benson D, Slichter SJ. Red cell collection by apheresis technology. Transfusion. 1993 Oct;33(10):819-24. doi: 10.1046/j.1537-2995.1993.331094054618.x. PMID 8236422
- [Background] Bolgiano DC, Smith S, Slichter SJ. Strategies to recruit plateletpheresis donors from a registry of HLA-typed, unrelated, bone marrow donors. Transfusion. 1993 Aug;33(8):675-8. doi: 10.1046/j.1537-2995.1993.33893342751.x. PMID 8342236